CLINICAL TRIAL: NCT04946175
Title: The Rate of Interventional Pain Procedures During Covid 19: A National Survey Among Egyptian Pain Practitioners
Brief Title: National Survey Among Egyptian Pain Practitioners
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ossama Hamdy Salman, Associate Professor, South Valley University
Other Study IDs: southvu8
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-05

CONDITIONS: Survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus pandemic health restrictions has deleteriously affected the rates of all interventional procedures even for emergency cases. This study tried to evaluate the impact of the outbreak of SARS-CoV-19 infection on rates of interventional pain therapy (IPT).

DETAILED DESCRIPTION:
Background: Coronavirus pandemic health restrictions has deleteriously affected the rates of all interventional procedures even for emergency cases. This study tried to evaluate the impact of the outbreak of SARS-CoV-19 infection on rates of interventional pain therapy (IPT).

Methods: Setting: Multicenter Study. Design: Prospective observational study, approved by the Local Ethical Committee (RC:2-1-21). Materials: Two 20-item questionnaires with five choices for probable answer using a Likert-5 point scale were constructed as self-assessment questionnaire. The questionnaires were uploaded to the Google drive, and the links and identification codes were sent using the WhatsApp to 500 IPT providers. The feedback answers were scored and statistically analyzed. Statistical analyses will be performed using IBM® SPSS® Statistics (Version 22, 2015; Armonk, USA) for Windows statistical package. P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

registered pain practitioners in Egypt.

-

Exclusion Criteria:

Non registered pain practitioners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: registered pain practitioners in Egypt.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
number of interventional pain procedures | June 1st 2020 till June 1st 2021
  questionnaire

SECONDARY OUTCOMES:
wearing protective clothing | june 1st 2020 to june 1st 2021
  during covid 19 pandemic

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - South Valley University Hospitals, Qina, Qena Governorate
  - South Valley University, Qina